CLINICAL TRIAL: NCT03757702
Title: Investigation of Trunk Position Sense, Postural Stability and Posture in Fibromyalgia Patients and Healthy Women
Brief Title: Trunk Position Sense, Postural Stability and Spinal Posture in Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 43
Record Dates: First submitted 2018-11-26; First posted 2018-11-29 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-11

CONDITIONS: Fibromyalgia; Postural Lordosis; Postural Kyphosis; Proprioception; Postural Stability; Balance
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromiyalgia group: women with FMS between 18-65 years of age and being volunteered.
  Interventions: Other: Evaluation
- Healthy group: healthy women and being volunteereed
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — Trunk position sense will be evaluated with a digital inclinometer. Trunk reposition test will be used in evaluation.The postural stability will be evaluated with a special balance device in eyes opened and closed position. Ellipse area (mm2) and perimeter (mm) parameters will be recorded.The angles of thoracal kyphosis and lumbar lordosis will be evaluated with a digital inclinometer.

SUMMARY:
This study aims to investigate trunk position sense, postural stability and spine posture in fibromyalgia patients and healthy women.

ELIGIBILITY:
Inclusion Criteria:

* being women
* having FMS
* being volunteer

Exclusion Criteria:

* have neurologic, infectious, endocrine, and other severe psychological disorders
* malignancy,
* being pregnant
* any condition interfering with evaluation (advanced cardiac respiratory or orthopedic problems)
* spinal deformities such as scoliosis, spine surgery
* inflammatory rheumatic diseases

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy women and Fibromyalgia patient
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Joint Position Sense | 20 days
  Trunk position sense will be evaluated with a digital inclinometer.

SECONDARY OUTCOMES:
Postural Stability | 20 days
  The postural stability will be evaluated with a special balance device in eyes opened and closed position.
Spinal Posture | 20 days
  .The angles of thoracal kyphosis and lumbar lordosis will be evaluated with a digital inclinometer.

CONTACTS AND LOCATIONS:
Overall Officials: Özge Çoban, Study Chair — Research Assitant
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No